CLINICAL TRIAL: NCT07173127
Title: The Effect of a Novel Combined Hormonal Treatment Containing a GnRH-antagonist for Uterine Fibroids and Endometriosis on Hemostasis Parameters: a Prospective Cohort Study
Brief Title: The Impact of a Novel GnRH Antagonist With Add-back Therapy for Treatment of Uterine Fibroids and Endometriosis on Hemostasis Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Manuela Viviano, MD, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-01609; 71434 (Other Grant/Funding Number: Hôpitaux Universitaires de Genève)
Record Dates: First submitted 2025-08-20; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Uterine Fibroid
Keywords: Uterine fibroids; Endometriosis; GnRh Antagonist; Hemostasis markers
MeSH Terms: conditions — Leiomyoma; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hemostasis markers dosage (Other)
  Interventions: Drug: Ryeqo treatment

INTERVENTIONS:
Drug: Ryeqo treatment — Ryeqo treatment will be administered and hemostasis markers will be measured at T0 and T1

SUMMARY:
Uterine fibroids and endometriosis are two frequent diseases among women of reproductive age. They can be responsible for chronic and/or menstrual pelvic pain and abnormal uterine bleeding. The first-line management of these conditions relies on medical treatment. Hormonal treatment with contraceptive pill can be effective, although up to 30% of patients do not respond to this line of treatment. In this context, GnRH antagonists have been introduced. By suppressing ovulation, they inhibit the action of the gonadal axis and thus can reduce bleeding and pain associated with uterine fibroids and endometriosis. More recently, the GnRH antagonist known as Relugolix has been associated with a low-dose oestradiol and progesteron-line molecule, a medication known as Ryeqo. The goal of this type of treatment is to suppress ovulation while also minimizing symptôms which may derive from lack of oestrogen and progesterone in reproductive age women.

While Ryeqo's efficacy has been proven by multiple large randomized controlled trials, its impact on blood coagulation has yet to be determined. Venous thromboembolism (VTE) is the main, potentially fatal, dleterious effect of oestrogen-containing hormonal treatmen, such as combined oral contraceptives (COC). Several epidemiological studies have found a 3-6 increase in the risk of VTE among women on COC. The thrombogenic risk can be assessed by measuring specific blood biomarkers, which are known to be correlated to the thrombogenic phenotype and allow an overview of the VTE risk prior to conducting large population-scale studies directly measuring the adverse event's prevalence.

The aim of this study is to document the effects of Ryeqo® on hemostasis parameters in order to estimate the risk of VTE associated with its employ. An improved understanding of the VTE risk associated with Ryeqo® will allow to adapt hormonal treatment based on each woman's personal risk profile.

The study will be explained to all women whose medical condition allows the prescription of Ryeqo. All women who give their consent to participate in the study will have a urinary pregnancy test and a blood sample drawn before beginning treatment with Ryeqo. A second visit will be scheduled at 3 months, throughout which a second blood sample will be drawn. A questionnaire including socio-demographic data and clinical symptoms will be completed both on the first and the second visit.

DETAILED DESCRIPTION:
Uterine fibroids, also known as myomas, are one of the most frequently observed hormonal-dependent benign tumours of the female genital tract. Their prevalence is estimated to be up to 68% among reproductive age women and they can be responsible for invalidating symptoms, such as abnormal uterine bleeding, pelvic pain, infertility and/or symptoms derived from pelvic compression. The treatment of uterine fibroids depends on their size, number, location and the patient's wish to preserve her uterus. It includes hormonal therapy (progestin-only, agonists or antagonists of the gonadotropin-releasing hormone [GnRH]), surgery (myomectomy or hysterectomy), thermal ablation through radiofrequencies or focalised ultrasounds and radiological uterine artery embolization.

Endometriosis is a chronic disease affecting 10% of reproductive age women. It can be responsible for symptoms such as pelvic pain in the form of dysmenorrhea, chronic pain and dyspareunia, as well as infertility. These symptoms depend on the proliferation of endometriotic lesions which, in turn, occurs mainly under the influence of oestradiol. Because of this physio-pathological mechanism, international guidelines recommend the use of medical treatment in order to lower oestradiol synthesis by inhibiting ovulation. Similarly to uterine fibroids, medical treatment includes oestro-progestin or progestin-only pill, agonists and antagonists of the GnRH.

As of February 2023, Swissmedic has approved the combined hormonal therapy known as Ryeqo® for treatment of abnormal uterine bleeding associated with uterine fibroids. Ryeqo® consists of an oral treatment, available as a pill, which contains 40 mg of the GnRH antagonist Relugolix, combined with 1 mg of oestradiol and a progestin, such as norethisterone acetate, at the dose of 0.5 mg. As the GnRH antagonist suppresses the hypothalamus-pituitary-gonadal axis, its combination with add -back hormonal replacement therapy maintains a low but constant oestradiol level, which minimizes vasomotor symptoms and long-term consequences of oestrogen deficiency, such as bone mineral density loss. Recent studies have assessed the efficacy of Ryeqo® for both abnormal uterine bleeding associated with uterine fibroids and endometriosis-associated pain, leading to the recent approval, as of April 2025, of Ryeqo® not only for uterine fibroids but also for treatment of moderate to severe pain among women with endometriosis in Switzerland.

While the efficacy of Ryeqo® in the management of abnormal uterine bleeding associated with uterine fibroids and pelvic pain due to endometriosis has been established, the drug's impact on hemostasis parameters has yet to be determined. This particular aspect merits attention, considering that the incidence of venous thromboembolism (VTE) varies based on age and is estimated to be 1-2/10,000 women-year between 15 and 34 years of age, and 3-5/10,000 women-year between 35 and 44 years of age. The clinical presentation varies between pulmonary embolism, which is potentially fatal, and veinous thrombosis. VTE has relevant short- and long-term morbidity, with a risk of 2-4% of chronic pulmonary hypertension and 3-10% of moderate-to-severe post-thrombotic syndrome.

VTE is the main, potentially fatal, deleterious effect of oestrogen-containing hormonal treatment, such as combined oral contraceptives (COC). Several epidemiological studies have found a 3-6 increase in the risk of VTE among women on COC. The thrombogenic risk can be assessed by measuring specific blood biomarkers, which are known to be correlated to the thrombogenic phenotype and allow an overview of the VTE risk prior to conducting large population-scale studies directly measuring the adverse event's prevalence. For contraceptive and hormone therapy, sensitivity of thrombin generation to the activated protein C (APC) pathway is a validated surrogate biomarker for estrogen-related VTE risk. Dosage of sex hormone-binding globulin (SHBG) also allow to assess VTE risk among COC users. These two biomarkers are used to assess VTE risk of new COC preparations.

Although no studies have yet specifically assessed the thrombogenic risk associated with the administration of Ryeqo®, a pooled analysis based on five prospective cohort studies concluded that oestradiol alone was associated with a decreased risk of VTE compared to ethynyl-oestradiol, while norethindrone acetate was associated with a risk comparable to that of oestrogens and progestins. The two active compounds combined with a GnRH antagonist, however, have not been studied for what concerns their impact on VTE risk. Based on the available literature, it is reasonable to presume that Ryeqo®'s administration has an impact on coagulation markers, thus explaining why the treatment is currently contraindicated in women who are experiencing, or have in the past experienced, venous or arterial thromboembolic events or who are at increased risk of such events due to their personal medical history. For this same reason, women are advised to suspend treatment with Ryeqo® in case the risk of VTE may be temporarily increased.

The aim of this study is to document the effects of Ryeqo® on hemostasis parameters in order to estimate the risk of VTE associated with its employ. An improved understanding of the VTE risk associated with Ryeqo® will allow to adapt hormonal treatment based on each woman's personal risk profile.

ELIGIBILITY:
Inclusion Criteria:

* Women consulting at the DFEA of the HUG, who are prescribed Ryeqo® for a qualified medical condition
* Age ≥ 18 years

Exclusion Criteria:

* Unable to speak and/or read French
* Having used either an oestro-progestin pill (oral, patch or vaginal ring) or oral estrogens in the past 3 months, or DMPA or nomegestrol acetate
* Women not having given their consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean value of normalized activated protein C resistance (nAPCsr) at 3 months of treatment with Ryeqo | At baseline and after 3 months of treatment
  Blood dosage of normalized activated protein C resistance (nAPCsr)

SECONDARY OUTCOMES:
Mean change from baseline to 3 months of treament in the value of sexual hormone-binding globulin (SHBG) | At baseline and after 3 months of treatment
  Mean value of SHBG as expressed in nmol/l units
Mean change from baseline to 3 months of treament in the value of normalized thrombomodulin sensitivity ratios (nTMSR) | At baseline and after 3 months of treatment
  Mean value of nTMSR as expressed as ratio
Mean change from baseline to 3 months of treament in the value of D-Dimers | At baseline and after 3 months of treatment
  Mean value of D-dimers as expressed with ng/ml units
Mean change from baseline to 3 months of treament in the value of thrombin generation markers | At baseline and after 3 months of treatment
  Mean value of thrombin generation markers, such as :
  thrombin generation markers
  * endogenous thrombin potential (ETP), expressed in nMxmin
  * peak value, expressed in nM
  * time to peak, expressed in min
  * lag time, expressed in min
Mean change from baseline to 3 months of treament in the value of antithrombin activity | At baseline and after 3 months of treatment
  Mean change in antithrombin activity, expressed as a percentage
Mean change from baseline to 3 months of treament in the value of Tissue factor pathway inhibitor (TFPI) | At baseline and after 3 months of treatment
  Mean change in the value of TFPI, as expressed in ng/ml
Mean change from baseline to 3 months of treament in the value of fibrinogen | At baseline and after 3 months of treatment
  Mean change in the value of fibrinogen, as expressed in g/l
Mean change from baseline to 3 months of treament in the value of free protein S | At baseline and after 3 months of treatment
  Mean change in the value of free protein S, expressed as a percentage
Mean change from baseline to 3 months of treament in the value of factor VIII concentration | At baseline and after 3 months of treatment
  Mean change in the value of factor VIII concentration, expressed as a percentage
Mean change from baseline to 3 months of treament in the value of thrombin-antithrombin-komplex (TAT) | At baseline and after 3 months of treatment
  Mean change in the value of TAT concentration, expressed in microgr/l

OTHER OUTCOMES:
Mean days of headache at 3 months of treatment | At 3 months of treatment
  Number of participants having headache and, if so, mean numberof days spent experiencing headache
Mean number of days with pelvic pain at 3 months of treatment | At 3 months of treatment
  Number of participants experiencing pelvic pain and, if so, mean number of days spent with pelvic pain
Mean difference from baseline on the Higham scale of bleeding at 3 months of treatment | At baseline and after 3 months of treatment
  There is no minimum or maximum value. A score inferior to 100 indicates normal flow, a score of 100 or more suggests heavy bleeding, and a score of 150 or more signifies heavy bleeding
Mean number of days of experiencing hot flush | After 3 months of treatment
  Number of participants experiecing hot flush and, if so, mean number of days spent experiecing hot flush

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Petignat, Prof, Study Director — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data will be shared upon request, in anonymous form.

REFERENCES:
- [Background] Hugon-Rodin J, Fontana P, Poncet A, Streuli I, Casini A, Blondon M. Longitudinal profile of estrogen-related thrombotic biomarkers after cessation of combined hormonal contraceptives. Blood. 2024 Jan 4;143(1):70-78. doi: 10.1182/blood.2023021717. PMID 37939264